CLINICAL TRIAL: NCT04934657
Title: The Second Affiliated Hospital of Zhejiang University, School of Medicine
Brief Title: Association of Perioperative Daily Steps and Postoperative Recovery Among Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0344
Record Dates: First submitted 2021-06-08; First posted 2021-06-22 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Recovery
Keywords: daily step, recovery, length of hospital stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal steps: patients in this group have normal preoperative step counts
  Interventions: Other: no intervention
- low steps: patients in this group have low preoperative step counts
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Walking is the most common, simple and convenient way of exercise with the lowest cost. Studies have shown that daily steps are related to important health outcomes such as cardiovascular events and all-cause mortality. Catrine et al. believe that daily steps can be used as a basic index to evaluate physical fitness. Many observational studies have found that postoperative daily steps collected by wearable devices or smart phones are related to length of hospital stay or even postoperative depression, which is suggested that the average daily steps may be an important index to predict the prognosis of patients.

So the investigators aim to explore the association between peri-operative average daily steps and postoperative recovery of patients scheduled for elective surgery.

DETAILED DESCRIPTION:
Patients scheduled to undergoing elective surgery including thoracic surgery ,abdominal surgery, primary hip replacement and radical mastectomy will be recruited.The exclusion criteria are as follows: With preoperative unconsciousness; Day surgery (planned length of stay < 1 day); Wheelchair, walking aid or crutch were used before operation; Unable to walk due to physical limitations; The collection time of preoperative steps was less than 1 week; The patient refused to participate.

After recruitment and screening , the investigators will ask the participants to wear a smart band to record data of their daily steps , in addition the investigators will collect the peri-operative data of these participants which includes their rehabilitations and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled to undergo elective surgery including thoracic surgery abdominal surgery, primary hip replacement and radical mastectomy ; Age≥18 ASA Ⅰ～Ⅲ Able to wear smart band

Exclusion Criteria:

With preoperative unconsciousness Day surgery (planned LOS < 1 day) Wheelchair, walking aid or crutch were used before operation Unable to walk due to physical limitations The collection time of preoperative steps was less than 1 week The patient refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the participants are adult patients scheduled to undergo elective surgery including thoracic surgery ,abdominal surgery, primary hip replacement and radical mastectomy.They will be asked to wear smart band to record their daily steps when they do the preoperative evaluation.
Sampling Method: Probability Sample
Enrollment: 487 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the length of hospital stay | within 7 days after operation or before discharge, whichever came first
  postoperative length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, MD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao Y, Wang Y, Liu Y, Yu Y, Wang X, Wang T, Zheng B, Yan M. Association of perioperative step count tracked by a wristband with surgical outcomes in minimally invasive lung cancer surgery: a prospective observational study. Front Med (Lausanne). 2025 Jul 29;12:1590327. doi: 10.3389/fmed.2025.1590327. eCollection 2025. PMID 40800130